CLINICAL TRIAL: NCT03270553
Title: A Phase 1, Open Label, Randomized, 2-Period, 2-Treatment, Crossover Study to Assess the Effect of Plazomicin on the Pharmacokinetics of Metformin in Healthy Subjects
Brief Title: A Study to Assess the Effect of Plazomicin on the Pharmacokinetics of Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ACHN-490-011
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — plazomicin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): In Period 1, subjects receive metformin alone; in Period 2, subjects receive metformin + plazomicin
  Interventions: Drug: plazomicin; Drug: metformin
- Sequence 2 (Experimental): In Period 1, subjects receive metformin + plazomicin; in Period 2, subjects receive metformin alone
  Interventions: Drug: plazomicin; Drug: metformin

INTERVENTIONS:
Drug: plazomicin — single intravenous dose
Drug: metformin — single oral dose

SUMMARY:
This is a single-center, Phase 1, open label, randomized, two-sequence, two-period, crossover study to evaluate the drug-drug interaction potential between plazomicin and metformin in healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Medically healthy, with no clinically significant medical history, physical examination findings, vital signs, or ECG findings

Key Exclusion Criteria:

* Estimated creatinine clearance <90 mL/min
* Use of tobacco- or nicotine-containing products
* History in the past 90 days of prior trauma to the outer or internal structures of the ear or tinnitus
* History or family history of vestibular disorder, chronic vertigo (sensation of spinning), chronic dizziness
* History of hearing loss or a family history of hearing loss, or a prior diagnosis of sensorineural hearing loss or Ménière's disease

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2017-10-07 (Actual); Study Completion 2017-10-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of metformin in plasma | 9 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 15 days
Change from baseline in vital signs post dose (temperature, pulse, respiration, blood pressure) | 8 days
Absolute values of and change from baseline in clinical laboratory values (hematology, serum chemistry, urine analysis) | 9 days
Pharmacokinetics of metformin in urine | 9 days
Pharmacokinetics of plazomicin in plasma | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Shyeilla Dhuria, Study Director — Achaogen, Inc.
Locations (1):
- Clinical Site, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Choi T, Komirenko AS, Riddle V, Kim A, Dhuria SV. No Effect of Plazomicin on the Pharmacokinetics of Metformin in Healthy Subjects. Clin Pharmacol Drug Dev. 2019 Aug;8(6):818-826. doi: 10.1002/cpdd.648. Epub 2019 Jan 3. PMID 30605260